CLINICAL TRIAL: NCT03296319
Title: Echocardiography Guided Fluid Resuscitation in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Esam, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Echocardiography guided fluid
Record Dates: First submitted 2017-08-27; First posted 2017-09-28 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Fluid Responsiveness; Echocardiography
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- echocardiography guided fluid resuscitation (Active Comparator)
  Interventions: Device: Echocardiography
- clinically guided fluid resuscitation (Experimental)
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Echocardiography — Echocardiography guided fluid administration

SUMMARY:
To compare between the impact of echocardiography guided fluid resuscitation and clinically guided fluid resuscitation on critically ill patients in hospital outcome.

DETAILED DESCRIPTION:
Resuscitation often requires the infusion of intravenous fluid in an effort to reverse organ dysfunction. The harms of inappropriate use of fluid are becoming increasingly apparent The question of whether the patient improves with fluid, additional vasopressors or inotropes can be difficult to answer. The gold standard for assessing fluid responsiveness to guide fluid administration in critically ill patients is to perform a fluid challenge. The rationale for volume expansion is to increase the cardiac output (CO) and oxygen delivery to ultimately improve tissue oxygenation. This involves the infusion of a specific amount of intravenous fluid to assess ventricular preload reserve and subsequent systemic haemodynamic effects. In a patient with acute hemodynamic instability, a fluid challenge will cause an increase in stroke volume, according to the Frank-Starling curve. This increase in stroke volume has a salutary effect because it improves tissue perfusion. In contrast, higher hydrostatic pressures in the vascular system predispose the patient to edema, organic dysfunction, and increased risk of in-hospital mortality.

Fluid responsiveness is conventionally defined as an increase of at least 10% to 15% in SV in response to a fluid challenge, which is a reflection of the limits of precision of the technology used.

Assessment of the response in flow to a fluid challenge can be guided with echocardiography. It is achieved by measuring left ventricular outflow tract velocity time integral (LVOT VTI) immediately before and after fluid challenge.

ELIGIBILITY:
Inclusion Criteria:

1- All Critical ill-patients with Acute Physiologic Assessment and Chronic Health Evaluation II score (APACHE II score)≥ 25

Exclusion Criteria:

1. Bad echocardiographic window
2. APACHE II score < 25.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
The impact of echocardiography guided fluid resuscitation | Baseline
  we will compare the results of fluid administration between two groups of patients with APACHE II score > 25: the first group using clinical sense only and the other group using transthoracic echocardiography including: The sample box of PW Doppler will be placed at thelevel of the aortic valve or within 1 cm of it, in the LVOT. Peak velocity variation of 12% before and after 250 cc normal saline challenge in adults predicts fluid responsiveness (12) and VTI variation is also predictive. The percentage variations in SV, VTI or peak velocity are calculated using the following equation: variations =100 x svmax-svmin/(svmax+svmin) x 0.5.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine, Assiut university, Asyut, Egypt

REFERENCES:
- [Result] Jonas MM, Tanser SJ. Lithium dilution measurement of cardiac output and arterial pulse waveform analysis: an indicator dilution calibrated beat-by-beat system for continuous estimation of cardiac output. Curr Opin Crit Care. 2002 Jun;8(3):257-61. doi: 10.1097/00075198-200206000-00010. PMID 12386506
- [Result] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Result] Boyd JH, Forbes J, Nakada TA, Walley KR, Russell JA. Fluid resuscitation in septic shock: a positive fluid balance and elevated central venous pressure are associated with increased mortality. Crit Care Med. 2011 Feb;39(2):259-65. doi: 10.1097/CCM.0b013e3181feeb15. PMID 20975548
- [Result] Squara P, Cecconi M, Rhodes A, Singer M, Chiche JD. Tracking changes in cardiac output: methodological considerations for the validation of monitoring devices. Intensive Care Med. 2009 Oct;35(10):1801-8. doi: 10.1007/s00134-009-1570-9. Epub 2009 Jul 11. PMID 19593546
- [Result] Cecconi M, Parsons AK, Rhodes A. What is a fluid challenge? Curr Opin Crit Care. 2011 Jun;17(3):290-5. doi: 10.1097/MCC.0b013e32834699cd. PMID 21508838
- [Result] Hofer CK, Cannesson M. Monitoring fluid responsiveness. Acta Anaesthesiol Taiwan. 2011 Jun;49(2):59-65. doi: 10.1016/j.aat.2011.05.001. Epub 2011 Jun 24. PMID 21729812
- [Result] Vincent JL. "Let's give some fluid and see what happens" versus the "mini-fluid challenge". Anesthesiology. 2011 Sep;115(3):455-6. doi: 10.1097/ALN.0b013e318229a521. No abstract available. PMID 21792055
- [Result] Frazee E, Kashani K. Fluid Management for Critically Ill Patients: A Review of the Current State of Fluid Therapy in the Intensive Care Unit. Kidney Dis (Basel). 2016 Jun;2(2):64-71. doi: 10.1159/000446265. Epub 2016 May 18. PMID 27536694
- [Result] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Result] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Result] Chen C, Kollef MH. Conservative fluid therapy in septic shock: an example of targeted therapeutic minimization. Crit Care. 2014 Aug 29;18(4):481. doi: 10.1186/s13054-014-0481-5. PMID 25185073
- [Result] Teboul JL, Monnet X. Prediction of volume responsiveness in critically ill patients with spontaneous breathing activity. Curr Opin Crit Care. 2008 Jun;14(3):334-9. doi: 10.1097/MCC.0b013e3282fd6e1e. PMID 18467896